CLINICAL TRIAL: NCT07065318
Title: Comparison of the Effects of Continuous Aerobic Exercise Training and High-Intensity Interval Exercise Training on ICF-Based Assessments in Lung Transplant Candidates
Brief Title: Lung Transplant Candidates: Effects of Aerobic vs. HIIT Training on ICF Assessments
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Ulaş Ar, Principal Investigator, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TABED-2-24-305
Record Dates: First submitted 2024-11-21; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Lung Transplantation
Keywords: lung transplant candidates; exercise training; high intensity interval training; aerobic exercise

STUDY DESIGN:
Intervention Model Description: There will be 2 groups in the study. Group 1 will do low volume high-intensity interval exercise training. Group 2 will receive moderate-intensity continuous aerobic exercise training.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LV-HIIT (Low-Volume High-Intensity Interval Training) (Experimental): The first randomly assigned group will perform 30 seconds of high-intensity exercise at 85-100% of their maximum workload, followed by 30 seconds of exercise at 40% of their maximum workload. This 30-second high-intensity exercise followed by 30 seconds of low-intensity exercise will be referred to as one cycle. A total of 20 cycles will be completed. Additionally, 2 minutes of low-intensity warm-up and cool-down exercises will be performed.
  Interventions: Behavioral: LV-HIIT (Low-Volume High-Intensity Interval Training); Device: Ergometer cycle
- MICT (Moderate-Intensity Continuous Training) (Active Comparator): The second group determined as a result of randomization will exercise for 20-30 minutes at 60-80% of maximum workload. Exercise volume (duration × %Wpeak) matched between groups.
  Interventions: Behavioral: MICT (Moderate-Intensity Continuous Training); Device: Ergometer cycle

INTERVENTIONS:
Behavioral: LV-HIIT (Low-Volume High-Intensity Interval Training) — 30-sec intervals at 85-100% peak workload, 30-sec rest at 40%, total 20-30 min.
  Arms: LV-HIIT (Low-Volume High-Intensity Interval Training)
Behavioral: MICT (Moderate-Intensity Continuous Training) — Continuous cycling at 60-80% peak workload for 20-30 min.
  Arms: MICT (Moderate-Intensity Continuous Training)
Device: Ergometer cycle — Electronically Ergometer cycle custo ec5000, CustoMed used for all exercise sessions. Calibrated before each trial.

SUMMARY:
Lung transplantation is a crucial surgical intervention aimed at increasing survival rates in patients with end-stage lung diseases such as chronic obstructive pulmonary disease (COPD), cystic fibrosis, idiopathic pulmonary fibrosis, and pulmonary hypertension. One of the most important determinants of health outcomes before and after lung transplantation is exercise capacity. An increase in the 6-minute walking distance (6MWD), which serves as a measure of functional exercise capacity, is associated with lower mortality rates in both pre- and post-transplantation settings. Therefore, effective rehabilitation programs are needed to enhance the exercise capacities of lung transplant candidates.

Pulmonary rehabilitation (PR) is a comprehensive program designed specifically for individuals with chronic respiratory diseases. PR aims to improve patients' physical and psychological conditions through detailed assessments and personalized treatment plans. It can play a role in enhancing the preoperative exercise capacities of lung transplant candidates and improving their chances of successful health outcomes. However, lung transplant candidates often have more advanced lung disease and face greater challenges compared to typical patients undergoing PR, making the expected benefits more complex to achieve.

The primary aim of this study is to investigate the effects of high-intensity interval training (HIIT) in lung transplant candidates with interstitial lung disease (ILD). The first objective is to compare the physiological responses and effectiveness of HIIT and moderate-intensity continuous training (MICT) within the same exercise volume. The secondary aim is to evaluate the impact of HIIT on body structure and function, activity, and participation levels using ICF-based assessments.

DETAILED DESCRIPTION:
Research Design This study employs a randomized controlled prospective design. The exercise training protocol consists of two main groups: high-intensity interval training (HIIT) and moderate-intensity continuous training (MICT). The HIIT protocol includes high-intensity efforts performed in 30-second intervals, while the MICT protocol involves longer-duration, moderate-intensity exercise. The total training duration for both groups is planned for 8 weeks.

Participants will include individuals with interstitial lung disease who are on the waiting list for lung transplantation. They must agree to participate regularly in the exercise program. Power analysis indicated that a minimum of 17 participants per group is needed, leading to a total target of 34 participants.

Parameters to be Assessed The study will assess various parameters before and after the exercise training. These parameters include demographic information, exercise capacity, respiratory function, comorbidities, daily living activities, and quality of life.

Exercise capacity will be evaluated using the 6-minute walk test (6MWT). Respiratory functions will be measured through pulmonary function tests (PFT), capturing values such as forced expiratory volume in one second (FEV1), forced vital capacity (FVC), and carbon monoxide diffusion capacity (DLCO). Comorbidities will be assessed using the Charlson Comorbidity Index, while daily living activities will be measured using the London Chest and St. George questionnaires.

Quality of life will be evaluated through various scales. For instance, the Tampa Kinesiophobia Scale will assess fear and anxiety levels in patients. Additionally, the FRAIL Scale will evaluate frailty, sarcopenia levels, and muscle strength.

Hypotheses

This study has four main hypotheses:

There is a significant difference between HIIT and MICT regarding the effects on body structure and function impairments, activity, and participation levels.

HIIT has a positive effect on respiratory function, exercise capacity, and quality of life.

HIIT has an effect on sarcopenia and frailty levels. HIIT impacts body structure and function impairments, activity, and participation levels.

Conclusion This study aims to evaluate the effects of high-intensity interval training in lung transplant candidates. The findings may contribute to optimizing pre-transplant rehabilitation processes and improving the overall health status of these patients. Furthermore, the applicability and effectiveness of such exercise protocols may lead to significant changes in clinical practice. The results of the research will shed light on the development of exercise rehabilitation programs and the treatment processes for lung disease patients.

ELIGIBILITY:
Inclusion Criteria:

* Being diagnosed with interstitial lung disease and being followed up at the Ankara City Hospital Chest Diseases Clinic,
* Being 18 years of age or older,
* Patients who are being followed up with a diagnosis of ILD according to the ATS/ERS 2022 international ILD guideline,
* Being on the lung transplant waiting list according to the International Society for Heart and Lung Transplantation and are being evaluated for listing and are being followed up by the chest diseases department (25-28),
* Being willing to participate in the exercise program regularly and volunteering to participate in the study,
* Patients who have dyspnea levels of 2 and above according to the Modified Medical Research Council dyspnea scale and are able to ambulate,
* Patients who receive long-term oxygen support will be included.

Exclusion Criteria:

* Patients with a history of exertional syncope,
* Patients in acute exacerbation,
* Patients with sarcoidosis,
* Patients with serious comorbidities that may limit exercise (e.g. musculoskeletal, neurological or cardiovascular problems) will not be included.
* Patients with an aortic aneurysm greater than 5.5 cm,
* Patients with cardiovascular impediments to exercise during cardiological evaluations prior to pulmonary rehabilitation

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — men and women
Enrollment: 34 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise capacity | through study completion, an average of 1 year
  Peak Work Rate (PWR) PWR is determined through a symptom-limited incremental bicycle ergometer test. Patients pedal at 10 W, increasing by 10 W each minute until fatigue or a workload of 50 W is reached, or a fatigue level of 9 on the modified Borg scale. Workload and heart rate are monitored, with maximum workload (Wpeak) and heart rate recorded at the end.
Submaximal exercise capacity | through study completion, an average of 1 year
  -Minute Walk Test (6MWT) The 6MWT assesses exercise capacity in a 30-meter corridor by measuring the distance walked. It evaluates oxygen saturation, heart rate, and dyspnea using the Borg scale before and after the test. Participants walk at their own pace and can pause or use oxygen as needed.

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 Second (FEV1) Measured by Spirometry (Liters) | through study completion, an average of 1 year
  FEV1 will be assessed via CosmedQuark PFT Q-Box, Italy following. Participants will perform ≥3 reproducible maneuvers; the highest value within 5% repeatability will be recorded and reported in liters. Values will be expressed as absolute liters and % predicted using equation.
Fragility | through study completion, an average of 1 year
  Frail Frailty Scale It is a scale that evaluates the patient's fatigue, resistance, mobility, weight loss and other diseases by questioning them. The FRAIL scale, which consists of 5 items, receives 0 or 1 points according to the answers given by the patients, and a total of 0 points is considered as non-frail, 1-2 points as pre-frail and >2 points as frail.
Life Quality | through study completion, an average of 1 year
  St George Quality of Life Questionnaire
  It is a scale that measures the quality of life specific to respiratory diseases. It consists of a total of 50 items, 8 of which question the patient's symptoms, 16 of which question the activities, and 26 of which question the effects of the disease. While evaluating the symptoms, the patient's level of shortness of breath, cough, and sputum respiratory discomfort are questioned. While evaluating the activity component, physical activities that cause shortness of breath or are restricted due to shortness of breath are questioned. While evaluating the effects of the disease, it includes factors such as work, occupation, keeping health under control, and discomfort during daily living activities. The 3 sections of the test are calculated separately and the total score is calculated. A score of 0 indicates normal, a score of 100 indicates maximum disability
Kinesiophobia | through study completion, an average of 1 year
  The Tampa Scale for Kinesiophobia (TSK) is a validated 17-item questionnaire assessing fear of movement and reinjury in chronic pain patients, scored on a 4-point Likert scale (1=strongly disagree to 4=strongly agree). Total scores range from 17 (no kinesiophobia) to 68 (severe kinesiophobia), with scores ≥38 indicating clinically significant fear that may impair recovery.
Muscle strength | through study completion, an average of 1 year
  Hand Grip Strength Jamar (Jamar®, California, USA) brand hand dynamometer, which is valid in clinical studies, will be used to measure hand grip strength.
Balance | through study completion, an average of 1 year
  Timed-up and Go Test Test is a test performed to evaluate dynamic balance and functional mobility. A standardized chair, stopwatch and 3 meters of walking space are needed. The test begins while sitting in a chair, the individual gets up with the start command, walks 3 meters at normal walking speed, turns back and sits on the chair. Test completion time is recorded for scoring. Those who complete it in more than 15 seconds are considered to have impairment in daily living activities.
Sarcopenia | through study completion, an average of 1 year
  SARC-F The SARC-F questionnaire is a self-reported screening tool for sarcopenia risk, based on five components: Strength, Assistance in walking, Rising from a chair, Climbing stairs, and Falls. It takes its name from the initials of the components. Each item is scored from 0 to 2, with a total score of ≥4 indicating a high risk. In this study, SARC-F will be used to assess sarcopenia risk at baseline and follow-up.
Respiratory muscle strength | through study completion, an average of 1 year
  Maximum Inspiratory Pressure (MIP) (cmH₂O) Maximum Expiratory Pressure (MEP) (cmH₂O)
Respiratory Muscle Endurance | through study completion, an average of 1 year
  This test will be conducted at 60% of MIP for 10 minutes, with respiratory frequency and duration recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice K Kılıc, Prof. Dr., Study Chair — Ankara City Hospital Bilkent; Ebru CK Calık Kutukcu, Prof. Dr., Study Director — Hacettepe University
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hume E, Ward L, Wilkinson M, Manifield J, Clark S, Vogiatzis I. Exercise training for lung transplant candidates and recipients: a systematic review. Eur Respir Rev. 2020 Oct 28;29(158):200053. doi: 10.1183/16000617.0053-2020. Print 2020 Dec 31. PMID 33115788